CLINICAL TRIAL: NCT01323075
Title: Pharmacodynamic Comparison of Truncal Blocks in Patients With or Without Metabolic Disease (Kidney Failure, Diabetes)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2010/PC-02; 2010-024519-15 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Renal Insufficiency; Diabetes
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Renal insufficiency group: Patients in this group have renal insufficiency as defined by a creatinine clearance of < 30 ml/min without dialysis. These patients do not have diabetes.
  Interventions: Procedure: Truncal block
- Diabetic group: These patients have diabetes, but not renal insufficiency.
  Interventions: Procedure: Truncal block
- Non-exposed group: These patients have neither a neurological nor a metabolic disease and a creatine clearance of > 90 ml/min
  Interventions: Procedure: Truncal block

INTERVENTIONS:
Procedure: Truncal block — Patients will have a truncal block during hand or wrist surgery.

SUMMARY:
The primary objective is to demonstrate a longer period of neurologic recovery from a sensory block assessed in each test group versus the group without metabolic disease.

ELIGIBILITY:
General Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 1 month of follow up
* The patient is scheduled for hand or wrist surgery

Inclusion Criteria for the "Renal Insufficiency" group

* Patient has renal insufficiency as defined by a creatine clearance of < 30ml/min without dialysis

Inclusion Criteria for the "Diabetes" group

* Patient has chronic hyperglycemia, either a fasting glycemia > 1.26 g/l (7mmol/l) for longer than 5 years and receiving an oral, well-adjusted (last HBA1c < 6.5%)), non-insulin, antidiabetic treatment

Inclusion Criteria for the "Non-exposed" group

* Patient without metabolic or neurologic disease, with creating clearance > 90ml/min

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* Patient weighs less than 50 kg
* Score ASA > 4
* contra indication for locoregional anesthesia
* Severe metabolic and / or decompensated renal disease, cardiac or pulmonary decompensation
* Associated peripheral neuropathy associated with diabetes or kidney disease
* Associated central neuropathy associated (eg MS ... narrow cervical canal)
* Patients with both renal failure and diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three patient populations schelduled for surgery on the hand or wrist. The three groups include (1) patients with no metabolic or neurologic disease history, (2) patients with renal insufficiency but not diabetes and (3) patients with diabetes but not renal insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

PRIMARY OUTCOMES:
The duration of sensory block in minutes. | Day 0 (per-op)
  The duration of the sensory block in minutes. The beginning of this term is defined by the end of the axillary block (last injection), and the end of this period is defined by the reappearance of sensitivity to touch in the area anesthetized.

SECONDARY OUTCOMES:
Time necessary for completion of axillary blocks (1 / 3 upper humerus)(min) | Day 0 (per-op)
Time necessary for installing sensory and motor block (min) | Day 0 (per-op)
  Time necessary for installing sensory and motor block (min): defined by the delay between the end of the block injection and the occurrence of insensitivity of blocked territories
Failure of the block: yes / no | Day 0 (per-op)
  Failure of the block: yes / no: defined by an absence of sensory block
Presence of paresthesia: yes / no | Day 0 (per-op)
Occurrence of neurological complications, yes/no | Day 0 (post-op)
  Neurological: occurrence of complications (paresthesia, paralysis, paresis ....) that persist (or not) until the final postoperative evaluation
Occurrence of neurological complications, yes/no | 1 month
  Occurrence of neurological complications (paresthesia, paralysis, paresis ....)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Hôpital Lapeyronnie CHU de Montpellier, Montpellier
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart

REFERENCES:
- [Result] Cuvillon P, Casier M, Demattei C, Bernard N, Boisson C, Vialles N, Lhermite J, Ripart J, Capdevila X. Comparison of axillary nerve block duration using mepivacaine in non-insulin diabetic or renal insufficiency patients: a controlled observational matched multicenter trial. Minerva Anestesiol. 2019 Feb;85(2):124-132. doi: 10.23736/S0375-9393.18.12322-4. Epub 2018 Mar 27. PMID 29589414